CLINICAL TRIAL: NCT04743388
Title: Study of the Kinetics of Antibodies Against SARS-CoV-2 and of Cellular Subpopulations of the Immune System in Volunteers Receiving the BNT162b2 Vaccine or Other Approved Vaccine Against SARS-CoV-2
Brief Title: Study of the Kinetics of Antibodies Against COVID-19 (SARS-CoV-2) and of Cellular Subpopulations of the Immune System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Prof Evangelos Terpos, Professor of Therapeutics-Hematology, National and Kapodistrian University of Athens
Other Study IDs: 900/24-12-2020
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: COVID-19; Healthy Volunteers; Chronic Disease; Hematological Malignancies; Solid Tumor
Keywords: COVID-19; BNT162b2 vaccine; Antibodies; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Chronic Disease; Hematologic Neoplasms | interventions — BNT162 Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — Blood samples (whole blood)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: Approximately 300 volunteers, healthy or with chronic diseases (diabetes mellitus, hypertension, heart disease, CRF, etc.) with no autoimmune disorders.
  Interventions: Biological: BNT162b2; Biological: Other vaccine against SARS-Cov-2
- Cohort 2: People with hematological malignancies or solid tumors in various phases of their treatment (under treatment or in remission/ follow-up). This cohort may include patients with smoldering multiple myeloma (n=50), multiple myeloma (n=140), chronic lymphocytic leukemia (with or without hypoglobulinemia) (n=50), lymphoma (n=80), AL amyloidosis (n=30), patients who receive PARP (n=30), CDK4/6 (n=30), or immune checkpoint inhibitors (n=40), and patients under therapy with Androgen Receptor Targeted Agents (n=50).
  Interventions: Biological: BNT162b2; Biological: Other vaccine against SARS-Cov-2

INTERVENTIONS:
Biological: BNT162b2 — Vaccine against SARS-Cov-2 of the Pfizer/BioNTech companies
Biological: Other vaccine against SARS-Cov-2 — Any other vaccine authorized and administered by the Greek Ministry of Health against SARS-Cov-2

SUMMARY:
Determination of both the degree and duration of the immunity provided after receiving the BNT162b2 vaccine against SARS-Cov-2.

DETAILED DESCRIPTION:
The purpose of this study is to assess the kinetics of antibodies against SARS-CoV-2 as well as the kinetics of the immune system's cell subpopulations and cytokines associated with the immune system in healthy volunteers receiving the BNT162b2 vaccine against SARS-Cov-2 of the Pfizer/BioNTech companies or any other vaccine authorized and administered by the Ministry of Health. Immunoassays will be performed at serum collection points before and after vaccination, as set out in this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers and all individuals who, according to the instructions of the Greek State are considered eligible to receive the BNT162b2 vaccine
* Age ≥ 18 years old

Exclusion Criteria:

* Serious allergy problems i.e. hospitalization due to a serious allergic reaction (anaphylaxis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The admission criteria include both healthy volunteers and all individuals who, according to the instructions of the Greek State are considered eligible to receive the BNT162b2 vaccine. In particular, the study includes people with hematological malignancies or solid tumors, either receiving treatment or in remission/ follow-up, pursuant to the vaccination instructions of the Ministry of Health. The study will also include patients with autoimmune diseases who receive or do not receive treatment for their disease. Patients with diabetes mellitus, hypertension, heart disease, chronic renal failure of all stages (and undergoing dialysis) or other chronic diseases deemed suitable for vaccination, according to the instructions of the Ministry of Health, may also participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Neutralizing antibodies against SARS-CoV-2 | Day 50 (28 days after the second dose of the vaccine)
  Primary endpoint of the study is the development of neutralizing antibodies against SARS-CoV-2 on Day 50 28 days after the second dose of the vaccine) in the study populations

SECONDARY OUTCOMES:
Neutralizing antibodies against SARS-CoV-2 | Day 1
  Development of neutralizing antibodies against SARS-CoV-2 on day 1 (before the first dose of the vaccine)
Neutralizing antibodies against SARS-CoV-2 | Day 8
  Development of neutralizing antibodies against SARS-CoV-2 on day 8
Neutralizing antibodies against SARS-CoV-2 | Day 22
  Development of neutralizing antibodies against SARS-CoV-2 on day 22 (before the second dose of the vaccine)
Neutralizing antibodies against SARS-CoV-2 | Day 36
  Development of neutralizing antibodies against SARS-CoV-2 on day 36
Neutralizing antibodies against SARS-CoV-2 | Month 3
  Development of neutralizing antibodies against SARS-CoV-2 at 3 months post the second dose of the vaccine
Neutralizing antibodies against SARS-CoV-2 | Month 6
  Development of neutralizing antibodies against SARS-CoV-2 at 6 months post the second dose of the vaccine
Neutralizing antibodies against SARS-CoV-2 | Month 9
  Development of neutralizing antibodies against SARS-CoV-2 at 9 months post the second dose of the vaccine
Neutralizing antibodies against SARS-CoV-2 | Month 12
  Development of neutralizing antibodies against SARS-CoV-2 at 12 months post the second dose of the vaccine
Neutralizing antibodies against SARS-CoV-2 | Month 18
  Development of neutralizing antibodies against SARS-CoV-2 at 18 months post the second dose of the vaccine
Development of anti-S-RBD antibodies against SARS-CoV-2 | Day 1
  Development of anti-S-RBD antibodies against SARS-CoV-2 on day 1 (before the first dose of the vaccine)
Development of anti-S-RBD antibodies against SARS-CoV-2 | Day 8
  Development of anti-S-RBD antibodies against SARS-CoV-2 on day 8
Development of anti-S-RBD antibodies against SARS-CoV-2 | Day 22
  Development of anti-S-RBD antibodies against SARS-CoV-2 on day 22 (before the second dose of the vaccine)
Development of anti-S-RBD antibodies against SARS-CoV-2 | Day 36
  Development of anti-S-RBD antibodies against SARS-CoV-2 on day 36
Development of anti-S-RBD antibodies against SARS-CoV-2 | Day 50
  Development of anti-S-RBD antibodies against SARS-CoV-2 on day 50
Development of anti-S-RBD antibodies against SARS-CoV-2 | Month 3
  Development of anti-S-RBD antibodies against SARS-CoV-2 at 3 months post the second dose of the vaccine
Development of anti-S-RBD antibodies against SARS-CoV-2 | Month 6
  Development of anti-S-RBD antibodies against SARS-CoV-2 at 6 months post the second dose of the vaccine
Development of anti-S-RBD antibodies against SARS-CoV-2 | Month 9
  Development of anti-S-RBD antibodies against SARS-CoV-2 at 9 months post the second dose of the vaccine
Development of anti-S-RBD antibodies against SARS-CoV-2 | Month 12
  Development of anti-S-RBD antibodies against SARS-CoV-2 at 12 months post the second dose of the vaccine
Development of anti-S-RBD antibodies against SARS-CoV-2 | Month 18
  Development of anti-S-RBD antibodies against SARS-CoV-2 at 18 months post the second dose of the vaccine
Number of memory B-cells against SARS-CoV-2 | Day 1
  According to antibody responses on day 1
Number of memory B-cells against SARS-CoV-2 | Day 8
  According to antibody responses on day 8
Number of memory B-cells against SARS-CoV-2 | Day 22
  According to antibody responses on day 22 (before the second dose of the vaccine)
Number of memory B-cells against SARS-CoV-2 | Day 36
  According to antibody responses on day 36
Number of memory B-cells against SARS-CoV-2 | Day 50
  According to antibody responses on day 50
Number of memory B-cells against SARS-CoV-2 | Month 3
  According to antibody responses at 3 months post the second dose of the vaccine
Number of memory B-cells against SARS-CoV-2 | Month 6
  According to antibody responses at 6 months post the second dose of the vaccine
Number of memory B-cells against SARS-CoV-2 | Month 9
  According to antibody responses at 9 months post the second dose of the vaccine
Number of memory B-cells against SARS-CoV-2 | Month 12
  According to antibody responses at 12 months post the second dose of the vaccine
Number of memory B-cells against SARS-CoV-2 | Month 18
  According to antibody responses at 18 months post the second dose of the vaccine
Number of memory T-cells against SARS-CoV-2 | Day 1
  According to antibody responses on day 1
Number of memory T-cells against SARS-CoV-2 | Day 8
  According to antibody responses on day 8
Number of memory T-cells against SARS-CoV-2 | Day 22
  According to antibody responses on day 22 (before the second dose of the vaccine)
Number of memory T-cells against SARS-CoV-2 | Day 36
  According to antibody responses on day 36
Number of memory T-cells against SARS-CoV-2 | Day 50
  According to antibody responses on day 50
Number of memory T-cells against SARS-CoV-2 | Month 3
  According to antibody responses at 3 months post the second dose of the vaccine
Number of memory T-cells against SARS-CoV-2 | Month 6
  According to antibody responses at 6 months post the second dose of the vaccine
Number of memory T-cells against SARS-CoV-2 | Month 9
  According to antibody responses at 9 months post the second dose of the vaccine
Number of memory T-cells against SARS-CoV-2 | Month 12
  According to antibody responses at 12 months post the second dose of the vaccine
Number of memory T-cells against SARS-CoV-2 | Month 18
  According to antibody responses at 18 months post the second dose of the vaccine
Number of monocytes (CD14+, CD16+) | Day 1
  According to antibody responses on day 1
Number of monocytes (CD14+, CD16+) | Day 8
  According to antibody responses on day 8
Number of monocytes (CD14+, CD16+) | Day 22
  According to antibody responses on day 22 (before the second dose of the vaccine)
Number of monocytes (CD14+, CD16+) | Day 36
  According to antibody responses on day 36
Number of monocytes (CD14+, CD16+) | Day 50
  According to antibody responses on day 50
Number of monocytes (CD14+, CD16+) | Month 3
  According to antibody responses at 3 months post the second dose of the vaccine
Number of monocytes (CD14+, CD16+) | Month 6
  According to antibody responses at 6 months post the second dose of the vaccine
Number of monocytes (CD14+, CD16+) | Month 9
  According to antibody responses at 9 months post the second dose of the vaccine
Number of monocytes (CD14+, CD16+) | Month 12
  According to antibody responses at 12 months post the second dose of the vaccine
Number of monocytes (CD14+, CD16+) | Month 18
  According to antibody responses at 18 months post the second dose of the vaccine
Interleukin 6 (IL-6), Interleukin 3 (IL-3), Interleukin 1b (IL-1b) levels | Day 1
  Inflammatory cytokines measurements on day 1 (before the first dose of the vaccine)
Interleukin 6 (IL-6), Interleukin 3 (IL-3), Interleukin 1b (IL-1b) levels | Day 8
  Inflammatory cytokines measurements on day 8
Interleukin 6 (IL-6), Interleukin 3 (IL-3), Interleukin 1b (IL-1b) levels | Day 22
  Inflammatory cytokines measurements on day 22 (before the second dose of the vaccine)
Interleukin 6 (IL-6), Interleukin 3 (IL-3), Interleukin 1b (IL-1b) levels | Day 23
  Inflammatory cytokines measurements on day 23
Interleukin 6 (IL-6), Interleukin 3 (IL-3), Interleukin 1b (IL-1b) levels | Day 36
  Inflammatory cytokines measurements on day 36
Interleukin 6 (IL-6), Interleukin 3 (IL-3), Interleukin 1b (IL-1b) levels | Day 50
  Inflammatory cytokines measurements on day 50
Interleukin 6 (IL-6), Interleukin 3 (IL-3), Interleukin 1b (IL-1b) levels | Month 3
  Inflammatory cytokines measurements at 3 months post the second dose of the vaccine
Interleukin 6 (IL-6), Interleukin 3 (IL-3), Interleukin 1b (IL-1b) levels | Month 6
  Inflammatory cytokines measurements at 6 months post the second dose of the vaccine
Interleukin 6 (IL-6), Interleukin 3 (IL-3), Interleukin 1b (IL-1b) levels | Month 9
  Inflammatory cytokines measurements at 9 months post the second dose of the vaccine
Interleukin 6 (IL-6), Interleukin 3 (IL-3), Interleukin 1b (IL-1b) levels | Month 12
  Inflammatory cytokines measurements at 12 months post the second dose of the vaccine
Interleukin 6 (IL-6), Interleukin 3 (IL-3), Interleukin 1b (IL-1b) levels | Month 18
  Inflammatory cytokines measurements at 18 months post the second dose of the vaccine
TNF-a levels | Day 1
  Inflammatory cytokines measurements on day 1 (before the first dose of the vaccine)
TNF-a levels | Day 8
  Inflammatory cytokines measurements on day 8
TNF-a levels | Day 22
  Inflammatory cytokines measurements on day 22 (before the second dose of the vaccine)
TNF-a levels | Day 23
  Inflammatory cytokines measurements on day 23
TNF-a levels | Day 36
  Inflammatory cytokines measurements on day 36
TNF-a levels | Day 50
  Inflammatory cytokines measurements on day 50
TNF-a levels | Month 3
  Inflammatory cytokines measurements at 3 months post the second dose of the vaccine
TNF-a levels | Month 6
  Inflammatory cytokines measurements at 6 months post the second dose of the vaccine
TNF-a levels | Month 9
  Inflammatory cytokines measurements at 9 months post the second dose of the vaccine
TNF-a levels | Month 12
  Inflammatory cytokines measurements at 12 months post the second dose of the vaccine
TNF-a levels | Month 18
  Inflammatory cytokines measurements at 18 months post the second dose of the vaccine
CRP levels | Day 1
  CRP blood level measurements on day 1 (before the first dose of the vaccine)
CRP levels | Day 8
  CRP blood level measurements on day 8
CRP levels | Day 22
  CRP blood level measurements on day 22 (before the second dose of the vaccine)
CRP levels | Day 23
  CRP blood level measurements on day 23
CRP levels | Day 36
  CRP blood level measurements on day 36
CRP levels | Day 50
  CRP blood level measurements on day 50
CRP levels | Month 3
  Inflammatory cytokines measurements at 3 months post the second dose of the vaccine
CRP levels | Month 6
  Inflammatory cytokines measurements at 6 months post the second dose of the vaccine
CRP levels | Month 9
  Inflammatory cytokines measurements at 9 months post the second dose of the vaccine
CRP levels | Month 12
  Inflammatory cytokines measurements at 12 months post the second dose of the vaccine
CRP levels | Month 18
  Inflammatory cytokines measurements at 18 months post the second dose of the vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Terpos, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- Department of Clinical Therapeutics, General Hospital of Athens ALEXANDRA, Athens, Greece

IPD SHARING:
Plan to Share IPD: No
At the end of the study, the results will be announced in medical conferences or medical journals.

REFERENCES:
- [Derived] Rosati M, Terpos E, Homan P, Bergamaschi C, Karaliota S, Ntanasis-Stathopoulos I, Devasundaram S, Bear J, Burns R, Bagratuni T, Trougakos IP, Dimopoulos MA, Pavlakis GN, Felber BK. Rapid transient and longer-lasting innate cytokine changes associated with adaptive immunity after repeated SARS-CoV-2 BNT162b2 mRNA vaccinations. Front Immunol. 2023 Nov 27;14:1292568. doi: 10.3389/fimmu.2023.1292568. eCollection 2023. PMID 38090597
- [Derived] Terpos E, Fotiou D, Karalis V, Ntanasis-Stathopoulos I, Sklirou AD, Gavriatopoulou M, Malandrakis P, Iconomidou VA, Kastritis E, Trougakos IP, Dimopoulos MA. SARS-CoV-2 humoral responses following booster BNT162b2 vaccination in patients with B-cell malignancies. Am J Hematol. 2022 Oct;97(10):1300-1308. doi: 10.1002/ajh.26669. Epub 2022 Aug 2. PMID 35871310
- [Derived] Dagla I, Iliou A, Benaki D, Gikas E, Mikros E, Bagratuni T, Kastritis E, Dimopoulos MA, Terpos E, Tsarbopoulos A. Plasma Metabolomic Alterations Induced by COVID-19 Vaccination Reveal Putative Biomarkers Reflecting the Immune Response. Cells. 2022 Apr 6;11(7):1241. doi: 10.3390/cells11071241. PMID 35406806
- [Derived] Gavriatopoulou M, Terpos E, Ntanasis-Stathopoulos I, Briasoulis A, Gumeni S, Malandrakis P, Fotiou D, Migkou M, Theodorakakou F, Eleutherakis-Papaiakovou E, Kanellias N, Kastritis E, Trougakos IP, Dimopoulos MA. Poor neutralizing antibody responses in 106 patients with WM after vaccination against SARS-CoV-2: a prospective study. Blood Adv. 2021 Nov 9;5(21):4398-4405. doi: 10.1182/bloodadvances.2021005444. PMID 34529762